CLINICAL TRIAL: NCT06768424
Title: Comparison of Minimally Invasive Surgical Therapy in Combination With Platelet Rich Fibrine and Guided Biofilm Therapy Combined With Platelet Rich Fibrine in the Treatment of Solitaire Intrabony Periodontal Defect A Prospective RCT.
Brief Title: Comparison of MIST With PRF and GBT With PRF in the Treatment of Intrabony Periodontal Defect. A Prospective RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Pal Nagy, associate professor, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OGYÉI/55689-5/2023
Record Dates: First submitted 2024-07-10; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Intrabony Periodontal Defect
Keywords: Guided biofilm terapy; Platelet Rich Fibrine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test 1 Guided biofilm therapy in combinaton with Platelet rich fibrine (Experimental): Non surgical treatment performed to clean and decontaminate the intrabony defect, and filled with PRF
  Interventions: Device: Guided biofilm therapy; Procedure: Platelet Rich Fibrin
- Test 2 Minimally invasive surgical therapy in combination with Platelet rich fibrine (Experimental): Surgical procedure: Minimal invasive surical approach Platelet rich fibrine chops is used in order to fill the intrabony gap.
  Interventions: Procedure: Platelet Rich Fibrin; Procedure: Minimally Invasive Surgical Technique
- Control group (Active Comparator): The control group patients are treated only with guided biofilm therapy alone
  Interventions: Device: Guided biofilm therapy

INTERVENTIONS:
Device: Guided biofilm therapy — Use of Airflow Plus powder subgingivally on teeth with deep periodeontal pockets
  Arms: Control group; Test 1 Guided biofilm therapy in combinaton with Platelet rich fibrine
Procedure: Platelet Rich Fibrin — Pack Platelet Rich Fibrin chops into the intrabony periodontla defect
  Arms: Test 1 Guided biofilm therapy in combinaton with Platelet rich fibrine; Test 2 Minimally invasive surgical therapy in combination with Platelet rich fibrine
Procedure: Minimally Invasive Surgical Technique — Periodontal intrabony defect is treated by minimally invasive surgical intervention
  Arms: Test 2 Minimally invasive surgical therapy in combination with Platelet rich fibrine

SUMMARY:
The aim is to evaluate in a prospective, randomized, controlled clinical study the healing of a MIST procedure combined with PRF, or GBT combined with PRF. Clinical, radiological evaluation of the regenerative surgical method and the GBT non-surgical therapy in solitaire deep intrabony periodontal defect.

DETAILED DESCRIPTION:
This clinical study aims to clinically and radiologically evaluate the healing response of the periodontal tissues in there is not opened flap design to access the intrabony defect test 1 group where The pre- surgically prepared Platelet Rich fibrine is added into the previously cleaned defect. In the test 2 group a minimally invasive surgical approach is used to access to the intrabony pocket. After opening a flap the same procedure is used to prepare PRF, and added into the pocket. The pockets in the control Group is only cleaned by guided biofilm therapy. Periodontal clinical parameters measured at baseline and at 6 months serves for secondary. After six months the healing is evaluated with a standardized X-ray holder. The primary outcome value is the delta clinical attachment level (gain or loss) The main interest is how the PRF influence the non-surgical healing. Does it any advance of flap opening procedure in comparison with the GBT, if PRF is used.

ELIGIBILITY:
Inclusion Criteria:

* solitaire intrabony periodontal defect at least 4 mm

Exclusion Criteria:

* Periodontitis with intrabony defect (Intrabony component ≥ 4mm, defect radiological angulation > 25°,
* The patient is able to comply with the study -related procedures (i.e. good level of oral hygiene, follow-up procedures).
* Patients must not be heavy smokers (<5 cigarettes/day).
* furcation involvement
* Full mouth plaque and bleeding scores (FMPS and FMBS) of <15% (O'Leary et al. 1972).
* The patient is able to fully understand the nature of the study, signed informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Intrabony fill | 6 months
  The change of the intrabony component compared to the initial intrabony defect depth (in percentage), which is measured on standardised individualised x-ray.

SECONDARY OUTCOMES:
PPD | 6 months
  Pocket probing depth measured clinically by calibrated periodontal probe (UNC 15)
GR | 6 months
  Gingival recession measured clinically by calibrated periodontal probe (UNC 15)
CAL | 6 months
  Clinical attachment level measured clinically by calibrated periodontal probe (UNC 15)

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University Department of Periodontology, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miron RJ, Moraschini V, Fujioka-Kobayashi M, Zhang Y, Kawase T, Cosgarea R, Jepsen S, Bishara M, Canullo L, Shirakata Y, Gruber R, Ferenc D, Calasans-Maia MD, Wang HL, Sculean A. Use of platelet-rich fibrin for the treatment of periodontal intrabony defects: a systematic review and meta-analysis. Clin Oral Investig. 2021 May;25(5):2461-2478. doi: 10.1007/s00784-021-03825-8. Epub 2021 Feb 20. PMID 33609186
- [Background] Patel GK, Gaekwad SS, Gujjari SK, S C VK. Platelet-Rich Fibrin in Regeneration of Intrabony Defects: A Randomized Controlled Trial. J Periodontol. 2017 Nov;88(11):1192-1199. doi: 10.1902/jop.2017.130710. Epub 2017 Aug 18. PMID 28820322
- [Background] Miron RJ, Fujioka-Kobayashi M, Bishara M, Zhang Y, Hernandez M, Choukroun J. Platelet-Rich Fibrin and Soft Tissue Wound Healing: A Systematic Review. Tissue Eng Part B Rev. 2017 Feb;23(1):83-99. doi: 10.1089/ten.TEB.2016.0233. Epub 2016 Oct 10. PMID 27672729
- [Background] Cortellini P, Cortellini S, Bonaccini D, Tonetti MS. Modified minimally invasive surgical technique in human intrabony defects with or without regenerative materials-10-year follow-up of a randomized clinical trial: Tooth retention, periodontitis recurrence, and costs. J Clin Periodontol. 2022 Jun;49(6):528-536. doi: 10.1111/jcpe.13627. Epub 2022 Apr 25. PMID 35415940